CLINICAL TRIAL: NCT00042926
Title: A Trial Of Lymphatic Mapping And Sentinel Node Lymphadenectomy For Patients With T1 or T2 Clinically N0 Oral Cavity Squamous Cell Carcinoma
Brief Title: Diagnostic Trial in Patients Who Are Undergoing Surgery for Early Stage Mouth Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ACOSOG-Z0360; CDR0000069485 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Immunohistochemistry; Sentinel Lymph Node Biopsy; Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiolymphoscintigraphy + surgery (Experimental): Patients undergo radiolymphoscintigraphy comprising technetium Tc 99m sulfur colloid to identify the sentinel lymph nodes (SNL). Within 18 hours after radiolymphoscintigraphy, patients undergo resection of the primary oral cavity tumor and radioguided sentinel lymphadenectomy and regional cervical lymphadenectomy. Lymph nodes are examined by hematoxylin and eosin (H&E) staining. If negative by H&E, lymph nodes are further analyzed by immunohistochemistry.
  Patients are followed at 30 days.
  Interventions: Other: immunohistochemistry staining method; Procedure: conventional surgery; Procedure: lymphangiography; Procedure: radionuclide imaging; Procedure: sentinel lymph node biopsy; Radiation: technetium Tc 99m sulfur colloid

INTERVENTIONS:
Other: immunohistochemistry staining method
Procedure: conventional surgery
Procedure: lymphangiography
Procedure: radionuclide imaging
Procedure: sentinel lymph node biopsy
Radiation: technetium Tc 99m sulfur colloid

SUMMARY:
RATIONALE: Diagnostic procedures to detect cancer cells in sentinel lymph nodes may help plan effective cancer treatment.

PURPOSE: Diagnostic trial to study the effectiveness of lymph node mapping and sentinel lymph node lymphadenectomy in patients who are undergoing surgery to remove early-stage cancer of the mouth.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether a negative hematoxylin and eosin finding from the lymphatic mapping and sentinel node lymphadenectomy procedure accurately predicts the negativity of the other cervical lymph nodes in patients with stage I or II squamous cell carcinoma of the oral cavity.
* Determine the extent and pattern of disease spread in the nodal bed in these patients.
* Obtain data on the use of immunohistochemistry to assess nodes in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be > 18 years of age.
2. Patient must have an ECOG/Zubrod performance status of < 2.
3. Patient must have a histologically confirmed primary T1 or T2 invasive OCSCCA that is > 6mm and < 4 cm in size. The primary tumor must be amenable to curative resection and must be diagnosed within 42 days prior to surgery.
4. Patient must be clinically stage N0 confirmed with a negative imaging study employing contrastenhanced CT scan (or MRI with gadolinium in patients with iodine allergy). Lymph nodes will be considered positive if:

   * Greater than 1.5 cm in size for levels I and II.
   * Greater than 1 cm in size for levels III, IV, V and VI.
   * If any lymph node exhibits central necrosis, irregular enhancement of a poorly defined or irregular capsular border.
   * Groups of three or more asymmetrically located LNs, with a minimal axial diameter of 8 mm or more, in the suspected tumor drainage area are present.
   * NOTE: All CT scans must be read by a neuroradiologist.
5. Patient must be medically fit for neck dissection.
6. Patient or the patient's legally acceptable representative must provide a signed and dated written informed consent prior to registration or any study-related procedures.
7. Female patient of childbearing potential must have negative serum pregnancy test within 30 daysprior to registration.
8. If the patient is a survivor of a prior cancer, ALL of the following criteria are met:

   1. Patient has undergone potentially curative therapy for all prior malignancies,
   2. No evidence of any prior malignancies for at least 5 years with no evidence of recurrence (except for effectively treated basal cell or squamous carcinoma of the skin, carcinoma in-situ of the cervix that has been effectively treated by surgery alone, or lobular carcinoma in-situ of the ipsilateral or contralateral breast treated by surgery alone),
   3. Patient is deemed by their treating physician to be at low risk for recurrence from prior malignancies.

Exclusion Criteria:

1. Patient received prior treatment to the cervical lymph nodes, including surgery or radiation therapy.
2. Patient experienced prior extensive trauma to the anterior cervical region of the neck.
3. Patient has lesions that cross the vermilion border involving lip skin.
4. Patient has had previous tumor resection involving the neck.
5. Patient has had injections of radioactive material for previous scans within 48 hours of the radiolymphoscintigraphy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2002-05; Primary Completion 2007-05 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Proportion of non-SLN(s) negative patients | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Civantos, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center

REFERENCES:
- [Result] Civantos FJ, Zitsch RP, Schuller DE, Agrawal A, Smith RB, Nason R, Petruzelli G, Gourin CG, Wong RJ, Ferris RL, El Naggar A, Ridge JA, Paniello RC, Owzar K, McCall L, Chepeha DB, Yarbrough WG, Myers JN. Sentinel lymph node biopsy accurately stages the regional lymph nodes for T1-T2 oral squamous cell carcinomas: results of a prospective multi-institutional trial. J Clin Oncol. 2010 Mar 10;28(8):1395-400. doi: 10.1200/JCO.2008.20.8777. Epub 2010 Feb 8. PMID 20142602